CLINICAL TRIAL: NCT01974219
Title: HIV-related Accelerated Aging of the Airway Epithelium
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1306013986; 5R01HL118857 (NIH)
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: HIV; COPD; Chronic Obstructive Pulmonary Disease; Smoking
Keywords: HIV; COPD; Chronic Obstructive Pulmonary Disease; Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, Cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy nonsmokers: Healthy nonsmokers
- Healthy smokers: Healthy smokers
- COPD smokers: COPD smokers

SUMMARY:
In cigarette smokers that are HIV+, one of the most common HIV-associated non-AIDS conditions is the accelerated development of chronic obstructive pulmonary disease (COPD), a disorder associated with significant morbidity and mortality. Based on the knowledge that COPD in smokers starts in the small airway epithelium, this study is focused on examining the hypothesis that the accelerated development of COPD associated with HIV infection results, in part, from an interaction of HIV directly on the small airway epithelium or through infection of cellular components of the immune system, with mediators released by these immune cells evoking premature biologic aging of the small airway epithelium. By identifying the early events in the pathogenesis of the HIV-associated accelerated COPD in smokers, we aim to identify biologic targets to which pharmacologic therapies could be addressed.

DETAILED DESCRIPTION:
While the epidemiologic data linking HIV infection to an increased risk for COPD is clear, the pathogenesis of the accelerated development of COPD in HIV infected smokers is not understood. We have focused on the SAE as the central target for the accelerated development of COPD in HIV infected smokers, as there is extensive data pointing to the SAE as the initial site of lung pathology in cigarette smokers and the small airways are the major site of airflow obstruction in COPD. Further, the emphysema associated with COPD begins in alveoli surrounding the SAE, and prior to the development of clinical evidence of lung disease, the SAE of smokers exhibit marked disordered biology, including changes in DNA methylation and gene expression, and disordered differentiation. Importantly, we have observed that HIV infection "ages" the SAE, with exaggerated shortening of SAE telomeres in individuals infected with HIV compared to HIV - smokers.

We propose that the early events in the pathogenesis of the accelerated development of COPD in smokers with HIV infection results from the premature biologic aging of the small airway epithelium (SAE) mediated by the effects of direct HIV infection of the SAE and/or through the interaction of HIV-infected T cells and/or alveolar macrophages (AM) with the SAE, resulting in the disordered biology of the SAE that is central to the pathogenesis of COPD.

In cigarette smokers that are HIV+, one of the most common HIV-associated non-AIDS conditions is the accelerated development of chronic obstructive pulmonary disease (COPD), a disorder associated with significant morbidity and mortality. Based on the knowledge that COPD in smokers starts in the SAE, this proposal is focused on examining the hypothesis that the accelerated development of COPD associated with HIV infection results, in part, from an interaction of HIV directly on the small airway epithelium or through infection of cellular components of the immune system, with mediators released by these immune cells evoking premature biologic aging of the small airway epithelium. By identifying the early events in the pathogenesis of the HIV-associated accelerated COPD in smokers, we aim to identify biologic targets to which pharmacologic therapies could be addressed.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY VOLUNTEER RESEARCH SUBJECTS

* All study subjects should be able to provide informed consent
* Males or females ages 18 years and older
* Must provide HIV informed consent

VOLUNTEER RESEARCH SUBJECTS WITH LUNG DISEASE

* Must provide informed consent
* Males and females age 18 years and older
* Lung disease proven by at least one of the following: symptoms consistent with pulmonary disease; (2) chest X-rays consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and/or (6) diseases of organs with known association with lung disease
* Must provide HIV informed consent

Exclusion Criteria:

HEALTHY VOLUNTEER RESEARCH SUBJECTS

* Individuals not deemed in good overall health by the investigator will not be accepted into the study.
* Habitual use of drugs and/or alcohol within the past six months (Acceptable: - Marijuana one time in three months; average of two alcoholic beverages per day; drug and/or alcohol abuse is defined as per the DSM-IV Substance Abuse Criteria).
* Individuals with history of chronic lung disease, including asthma or with recurrent or recent (within three months) acute pulmonary disease will not be accepted into the study.
* Individuals with allergies to atropine or any local anesthetic will not be accepted into the study.
* Individuals with allergies to pilocarpine, isoproterenol, terbutaline, atropine or aminophylline will not be accepted into the study.
* Females who are pregnant or nursing will not be accepted into the study

VOLUNTEER RESEARCH SUBJECTS WITH LUNG DISEASE

* Any history of allergies to xylocaine, lidocaine, versed, valium, atropine, pilocarpine, isoproterenol, terbutaline, aminophylline, or any local anesthetic will not be included in the study.
* Habitual use of drugs and/or alcohol within the past six months (Acceptable: Marijuana one time in three months; average of two alcoholic beverages per day; drug and/or alcohol abuse is defined as per the DSM-IV Substance Abuse Criteria)
* Females who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New York Metropolitan area residents
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2013-12-23 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Gene expression changes in airway epithelium | One Year
  We examine the pathogenesis of the accelerated development of COPD in smokers with HIV infection and the premature biologic aging of the small airway epithelium (SAE) mediated by the effects of direct HIV infection of the SAE and/or through the interaction of HIV-infected T cells and/or alveolar macrophages (AM) with the SAE, resulting in the disordered biology of the SAE that is central to the pathogenesis of COPD.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College and Weill Cornell Medical Center, Department of Genetic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided